CLINICAL TRIAL: NCT02508181
Title: Intra Ocular Pressure After I-gel and Supreme Insertion
Brief Title: Comparison of Intra Ocular Pressure After Insertion of the LMA Supreme and LMA Proseal in Pediatric Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KOU KAEK 2015/14
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Intra Ocular Pressure
Keywords: intra ocular pressure; I-gel; LMA Supreme; strabismus surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I-gel intra ocular pressure (Active Comparator): supraglottic airway device
  Interventions: Device: I-gel
- LMA Supreme intra ocular pressure (Active Comparator): supraglottic airway device
  Interventions: Device: LMA Supreme

INTERVENTIONS:
Device: I-gel — supraglottic airway device without cuff
  Arms: I-gel intra ocular pressure
Device: LMA Supreme — supraglottic airway device with cuff
  Arms: LMA Supreme intra ocular pressure

SUMMARY:
The investigators enrolled pediatric patients who are undergoing strabismus surgery. The investigators insert either an I-gel or laryngeal mask airway Supreme and measure the intraocular pressures.

DETAILED DESCRIPTION:
We already know that tracheal intubation increased intraocular pressure. We tried to evaluate the change of the intra ocular pressure increase before, during and after insertion the I-gel and LMA Supreme supraglottic airway devices. We enrolled the pediatric patients who are undergoing to strabismus surgery.

ELIGIBILITY:
Inclusion Criteria:

* pediatrics > 2 years
* pediatrics < 7 years
* undergoing strabismus surgery

Exclusion Criteria:

* pediatrics < 2 years
* pediatrics > 7 years
* neuromuscular blockage using

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
intra ocular pressure | 15 minutes
  measurement the intra ocular pressure before, during and after insertion of the device

SECONDARY OUTCOMES:
vomiting | 2 hour
bradicardia | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University School of Medicine, Kocaeli, Turkey (Türkiye)